CLINICAL TRIAL: NCT04371484
Title: Proposal of a Method Using the PMSI and SNIIRAM National Databases to Estimate the Frequency of Physical Abuse and to Identify th Eassociated At-risk Situations and Consequences in Children Aged 0 to 5 Years in France
Acronym: MENFIS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: GILARD-PIOC AOI 2017
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-04

CONDITIONS: Child Abuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- children from 0 to 5 years old, hospitalized
  Interventions: Other: ICD-10

INTERVENTIONS:
Other: ICD-10 — A collection of ICD-10 codes used within the PMSI that relate to physical abuse.

SUMMARY:
The epidemiological data currently available on child abuse in France are very inadequate. They do not make it possible to know the number of child victims, nor the precise context and impact of this violence. Very often, the figures put forward are underestimated. Improving the knowledge of these situations would make it possible to develop targeted primary and secondary prevention programs. In this study, is proposed an innovative method of exploiting existing national databases, the PMSI and SNIIRAM, with the aim of 1) approaching an order of magnitude of the frequency of physical abuse in children and 2) evaluating its contexts and consequences. The PMSI is a high-quality database that has been used for many years for medical research purposes. It provides a large amount of epidemiological information and can be used to create cohorts large enough to detect rare events. The SNIIRAM/EGB data allows the recovery of all data on reimbursed consumption, such as drug treatments, biological examinations carried out or consultations (with general practitioners or specialists).

ELIGIBILITY:
Inclusion Criteria:

* All children aged 0 to 5 years hospitalized in France between 2007 and 2014.
* Based on ICD-10 codes generated within the PMSI, 3 groups of children were defined:

  1. those with at least one code dedicated to physical abuse,
  2. those with at least one code or "combination of codes" suspected of physical abuse, and
  3. all other hospitalized children, control group.

Exclusion Criteria: NA

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children hospitalized in France between 2007 and 2014
Sampling Method: Non-Probability Sample
Enrollment: 4002359 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
The number of confirmed diagnoses for child abuse | Through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France